CLINICAL TRIAL: NCT02295488
Title: Determinism of the Mechanism of Action of Specific Immunotherapy in Hymenoptera Venom Allergy
Acronym: MAISAVEN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2014/069/HP
Record Dates: First submitted 2014-10-21; First posted 2014-11-20 (Estimated); Last update posted 2019-10-25 (Actual); Status verified 2019-10

CONDITIONS: Hymenoptera Allergy
Keywords: hymenoptera puncture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Desensitization (Experimental): Blood intake for biological sampling during validated desensitization protocol (Alyostall®)
  Interventions: Procedure: biological sampling; Biological: Desensitization protocol (Alyostall®)

INTERVENTIONS:
Procedure: biological sampling — blood intake for biological sampling during validated desensitization protocol (Alyostall®)
Biological: Desensitization protocol (Alyostall®) — Validated desensitization protocol using Alyostall® performed

SUMMARY:
Currently, most of the protocols used for desensitization to Hymenoptera venoms consist of a very rapid increase in doses of venom extracts administered during the SIT in a day without systemic reaction of the patient which is not yet explained. The hypothesis is that this good tolerance is due to a rapid decrease in the response of mast cells and basophils to the allergen..

The main objective is to study basophil activation in response to the allergen during the first day of desensitization, measured by basophil activation test.

The initiation of desensitization follow a protocol of rapid growth rates. The basophil activation level in the course of desensitization will be analyzed by flow cytometry after in vitro stimulation by allergen.

Changes in T cell polarization is also analyzed by flow cytometry. Evolution of the expression of different proteins in blood basophils will be studied by measuring their messenger RNAs

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years and below 75 years age
* Patient who presented a generalized allergic reaction after an puncture of a hymenoptera
* Patient with positive skin tests against the venom of a hymenoptera
* Patient with positive specific IgE against the venom of a hymenoptera • to which an indication of accelerated desensitization was chosen in day hospitalization
* Information and consent signed by the patient
* Patient affiliated to french social security system
* For women of childbearing age, taking an effective contraceptive.

Exclusion Criteria:

* Patients with the following diseases: Mastocytosis, systemic infection or hospitalization within 4 weeks before inclusion, chronic inflammatory disease, cancer, unbalanced asthma, immune deficiency
* Patients on beta-blocker, following another specific immunotherapy, or ongoing immunosuppressive therapy.
* Pregnant or lactating
* People placed under judicial protection
* Patient participating or having participated in another biomedical research within six months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2015-03-23 (Actual); Primary Completion 2018-04-12 (Actual); Study Completion 2018-04-12 (Actual)

PRIMARY OUTCOMES:
Evolution of basophil activation test value | Day 1 - 3h30
  Evolution of the basophil activation test (% of activated basophils) between the morning before the start of desensitization (Alyostall®) and before the last dose of the first day

SECONDARY OUTCOMES:
Correlation between results of activation basophil test results and tolerance | Day 1 - 5h30
  Looking for a correlation between the results of activation basophil test (% of activated basophils) and tolerance on the one hand and on the other hand the effectiveness of clinically evaluated desensitization (Alyostall®)
Evolution of basophil surface markers | Day 1 - 5h30
  Evolution of activated basophil surface markers by cytometric flow (% of activated) between the start of desensitization and before the last injection of the fist day of desensitization (Alyostall®)

CONTACTS AND LOCATIONS:
Overall Officials: Luc THIBERVILLE, Pr, Principal Investigator — UH Rouen
Locations (1):
- Rouen University Hospital, Rouen, France